CLINICAL TRIAL: NCT02201134
Title: SEVOflurane Inhalation in CARdiac Arrest Resuscitated Patients Treated With Therapeutic Hypothermia
Acronym: SEVOCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other); Hopital Gabriel Montpied (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0199; 2014-001196-31
Record Dates: First submitted 2014-07-16; First posted 2014-07-25 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Arrest; Therapeutic Hypothermia
Keywords: Cardiac arrest; Therapeutic hypothermia; Sevoflurane; Sedation; Patient resuscitated from cardiac arrest; Requiring sedation; Adult patients; Patient covered by french health care system
MeSH Terms: conditions — Heart Arrest | interventions — Sevoflurane

ARMS (1):
- sevoflurane (Other)
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: sevoflurane

SUMMARY:
Studying the feasibility of an initial sedation with inhalated sevoflurane during therapeutic hypothermia of cardiac arrests resuscitated patients.

DETAILED DESCRIPTION:
Prospective clinical study in ICU with ventilated patients sedated with sevoflurane using the Mirus® and Anaconda® , establishing the feasibility of an initial sedation of patients resuscitated from cardiac arrest and treated with therapeutic hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* -Adult patients ventilated requiring therapeutic hypothermia in ICU
* Stable respiratory and hemodynamic conditions
* Epinephrine and norepinephrine infusion rate < 1,5 g/kg/min
* Consent of patients or family
* Arterial line
* Patients resuscitated after cardiac arrest
* No Flow < 10 min
* Low Flow < 20 min
* Neutropenia < 1 G/L
* Post traumatic cardiac arrest
* Contraindication of halogenated anesthesics
* Extra corporeal life support or intra aortic balloon pump

Exclusion Criteria:

* -Pregnant woman
* Hemodynamic instability
* Brain death defined by the disappearance of brain stem reflexes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Determination of the feasibility of a sedation with inhalated sevoflurane in cardiac arrest resuscitated patients | at day 1
  The feasibility is evaluated by the number of side effects due to treatment until discharge from hospital.

SECONDARY OUTCOMES:
Determination of neurological prognostic of patients at ICU and hospital discharge | at day 1
Determination of systemic complications and organ failures during hospitalisation | at day 1
Evaluation of systemic inflammation and evolution with cytokines | at day 1
Evaluation of markers specific of brain ischemia (S100 protein and neuron-specific enolase) | at day 1
  at 3 times: before starting sevoflurane sedation, 24 hours, 48 hours and 72 hours after starting sevoflurane sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France